CLINICAL TRIAL: NCT02436499
Title: Chronic Migraine Treatment With Botulinum Toxin-A: an Investigation of Functional Magnetic Resonance Imaging Changes."
Brief Title: Chronic Migraine Treatment With Botulinum Toxin-A: an Investigation of Functional Magnetic Resonance Imaging Changes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Dr. Behzad Mansouri (Co-Primary Investigator) (Unknown)
Responsible Party: Principal Investigator, Dr. Dana Turcotte, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2015:022
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Botox and fMRI screening (Experimental): Following baseline screening, participants will receive two subsequent treatments with botulinum-A toxin, each separated by 12 weeks. Participants will receive standardized botulinum-A toxin dosing for chronic migraine prophylaxis, comprised of 155 total units given at 31 specified sites across 7 head/neck muscles (protocol to be explicitly described in full protocol). Second dose of botulinum-A toxin will either be maintained at 155 total units as dosed initially, or be increased to 195 total units, depending on response to clinical questionnaires and examination to evaluate response and efficacy (to be described in full protocol, consistent with the "Follow-the-Pain Injection Paradigm").
  Interventions: Drug: Botulinum Toxin-A

INTERVENTIONS:
Drug: Botulinum Toxin-A
  Other Names: Botox

SUMMARY:
Pilot study evaluating effect of Botox injection treatment for 12 individuals suffering from chronic migraine on function MRI imaging, before and after treatment.

DETAILED DESCRIPTION:
A proposed 12 patients will be recruited for participation in the pilot study. Consenting patients between the ages of 18-65 years old with confirmed chronic migraine (as defined by International Headache Society criteria) and meeting all other inclusion criteria (to be described in full protocol) will be enrolled for participation in the trial. Participants currently receiving migraine prophylaxis will be tapered off the specified medication (tapering regimen to be determined by clinicians) and a 4-week washout period will be observed prior to baseline assessments and Botox treatment. These patients will be permitted to use acute migraine medications as required. Participants will undergo baseline migraine significance assessments, which will include Headache Impact Test (HIT-6), the Migraine Disability Assessment (MIDAS) questionnaire and the Migraine Impact Questionnaire. Baseline neurological assessment will also be conducted at this visit. Additionally, baseline Beck Depression and Anxiety Inventories will be completed.

Participants will also undergo baseline fMRI on the 3Tesla Siemens MRI magnet at the National Research Council (NRC) Building located at 435 Ellice Avenue in Winnipeg, Manitoba. At this time, both structural and resting state fMRI data will be acquired. A 72-hour minimum migraine-free period will be ensured before each individual is allowed to proceed with imaging. A localizer image will be obtained. This is used for determining the participant's head position and for setting up the field of view for all subsequent images. Next, a high-resolution 3-dimensional image will be taken of the whole brain. This will be acquired with the following imaging parameters [Siemens MP-RAGE sequence, 1mm thick slices, zero spacing between slices, repetition time of 1900 ms, echo time of 2.2 ms, in plane resolution of 0.94 x 0.94, 256 x 256 matrix size with a 24 cm field of view, 176 volumes, resulting in a 8 minute 6 second scan time]. After the high-resolution image has been acquired, the resting state fMRI data will be acquired with the following parameters [Siemens echo planar imaging (EPI) sequence, 3 mm thick slices, zero spacing between slices, repetition time of 3000 ms, echo time of 30 ms, flip angle of 90°, 64 x 64 matrix size, 24 cm field of view, 140 volumes, resulting in a 7 minute 9 second scan time]. This provides the data set for the functional connectivity analysis. The high-resolution anatomical data serves as the background for the display of the superimposed resting state fMRI data. All image data will be acquired with an alpha-numeric code representing the study protocol number and participant number; the data will be transferred to a flash drive and copied to the principal investigator's hard drive for analysis. All participant paperwork and data back-up will be securely stored in the principal investigator's locked filing cabinet.

Following baseline screening, participants will receive two subsequent treatments with botulinum-A toxin, each separated by 12 weeks. Participants will receive standardized botulinum-A toxin dosing for chronic migraine prophylaxis, comprised of 155 total units given at 31 specified sites across 7 head/neck muscles (protocol to be explicitly described in full protocol). Second dose of botulinum-A toxin will either be maintained at 155 total units as dosed initially, or be increased to 195 total units, depending on response to clinical questionnaires and examination to evaluate response and efficacy (to be described in full protocol, consistent with the "Follow-the-Pain Injection Paradigm"). Following initial treatment (Day=0) participants will be requested to maintain daily headache diaries, in which they will be asked to record symptoms of active migraine as well as the use of acute migraine medications on a daily basis, in order to track migraine frequency and severity (example of headache diary will be included in full protocol). Participant timeline will be as follows: Day 0 (baseline assessments, fMRI and first Botox injection), Day 28 (clinic follow-up), Day 56 (second fMRI), Day 84 (clinic follow-up and second injection), Day 112 (clinic follow-up) and Day 140 (third fMRI). Clinic follow-up will be scheduled for Days 28, 84 and 112 at which time adverse events will be reviewed, as well as headache frequency reported in daily headache diaries. At these time points, participants will also repeat the same assessments completed at the baseline visit, including the HIT-6, MIDAS and Migraine Impact Questionnaire. At study termination (Day=140) patients will undergo a final fMRI scan as per baseline MRI protocol previously described.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, 18-65 years of age with confirmed chronic migraine (defined as migraine headache with or without aura, occurring on > 15 days of each month for at least 3 months
* Headaches must have at least two of the following characteristics: unilateral location, pulsating quality, moderate-severe pain intensity and/or aggravation by or causing avoidance of routine physical activity (eg. Walking or climbing stairs)
* Headaches must also have at least one of: nausea and/or vomiting or photophobia and/or phonophobia.
* Patients must be cognitively able to understand questionnaires and be able to complete Headache Logs.
* Patients must be physically able to undergo treatment administration, including the required positional changes needed for administration.

Exclusion Criteria:

* Headaches that could be attributed to other causes, as determined by clinician, including medication overuse headaches and chronic tension type headache.
* Females of childbearing age with confirmed or suspected pregnancy, those planning on conceiving during the trial duration and women who are breastfeeding.
* Previous treatment with botulinum toxin-A for chronic migraine.
* Confirmed allergy to botulinum toxin-A or any of the product components.
* Contraindications to fMRI procedure.
* Patients unable to discontinue migraine prophylaxis medications, including tricyclic antidepressants, beta-blockers and various antiepileptic medications, either due to unwillingness or safety issues (eg. Antiepileptics being used to manage seizure disorder). This will be determined by clinician.
* Participants exhibiting severe depression (BDI score >40) and/or suicidal ideation. These individuals will receive appropriate medical follow-up for psychological management.
* Active skin infection at planned injection site(s).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
function MRI imaging changes | 140 days
  3 fMRI scans will be done - one prior to treatment and two subsequent scans at Day 56 and Day 140

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada